CLINICAL TRIAL: NCT00980681
Title: Evaluation of Dotarem-enhanced Magnetic Resonance Angiography (MRA) Compared to Time-Of-Flight (TOF) MRA in the Diagnosis of Renal Arterial Disease
Brief Title: Renal Magnetic Resonance Angiography (MRA) Study Comparing Dotarem and Time-Of-Flight (TOF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment.
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DGD-44-047
Record Dates: First submitted 2009-09-17; First posted 2009-09-21 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-04

CONDITIONS: Renal Disease
Keywords: Renal disease; Contrast agent; MRA
MeSH Terms: conditions — Kidney Diseases | interventions — gadoterate meglumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dotarem (Experimental): Each subject will receive one injection of Dotarem 0.2ml/kg.
  Interventions: Drug: Dotarem
- Time Of Flight (Other): Each subject will undergo a TOF Magnetic Resonance Angiography
  Interventions: Other: Time of Flight

INTERVENTIONS:
Drug: Dotarem — Each subject will receive one injection of Dotarem 0.2ml/kg
  Other Names: gadoteric acid, gadoterate meglumine
  Arms: Dotarem
Other: Time of Flight — Each subject will undergo a TOF MRA
  Arms: Time Of Flight

SUMMARY:
The study will evaluate the efficacy and safety of Dotarem enhanced MRA compared to TOF MRA in patients suffering from renal arterial disease.

DETAILED DESCRIPTION:
Each participant will undergo first a TOF MRA followed by a Dotarem-enhanced MRA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged more than 18 years
* Strongly suspected of having renal arterial disease
* Scheduled (or to be scheduled) to undergo arterial catheter-based X-ray angiography examination

Exclusion Criteria:

* Known grade IV or V chronic kidney disease (GFR<30 mL/min/1.73m²)
* Contraindication to MRI
* Acute renal dysfunction within the 6 months preceding Dotarem®-enhanced MRA examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DESCHE, MD, Study Director — Guerbet
Locations (1):
- Guerbet LLC, Bloomington, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started in Sept 2009 and stopped in February 2010. Radiology departments from hospital or private practices were participating.
Pre-assignment Details: Out of the 13 enrolled patients, three did not receive treatment, mainly due to the Sponsor decision to interrupt the study
Groups:
- TOF Followed by Dotarem-enhanced MRA: Each patient will undergo a Time-OF-Flight (TOF) Magnetic Resonance Angiography (MRA) followed by a Dotarem-enhanced MRA (with one injection of Dotarem 0.2ml/kg).
Period: TOF MRA
Arm/Group | TOF Followed by Dotarem-enhanced MRA
Started | 10 (Out of the 13 enrolled patients, three did not receive treatment)
Completed | 10
Not Completed | 0
Period: Dotarem MRA
Arm/Group | TOF Followed by Dotarem-enhanced MRA
Started | 10 (Out of the 13 enrolled patients, three did not receive treatment)
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TOF Followed by Dotarem-enhanced MRA
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 7
  Canada | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent of Non Assessable Renal Artery Segments
Description: For each examination (TOF and Dotarem-enhanced MRA) the percent of non-assessable segments will be compared
Time Frame: 1 to 7 days
Measure: Number; unit: percentage of non-assessable segments
Groups:
- Dotarem-enhanced MRA: Patients benefiting from an MRA after administration with Dotarem
- Time-Of-Flight MRA: Patients benefiting from an MRA with no injection of contrast medium
Arm/Group | Dotarem-enhanced MRA | Time-Of-Flight MRA
Number analyzed (Participants) | 10 | 10
percentage of non-assessable segments | 25 | 20

ADVERSE EVENTS:
Arm/Group | Dotarem | Time Of Flight
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dotarem (N=10) | Time Of Flight (N=10)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was not completed due to poor enrolment. The statistical analysis was not perfomed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days